CLINICAL TRIAL: NCT03912402
Title: Multicenter Open-Label Single-Arm Trial of the Efficacy and Safety of BCD-100 in Combination With Platinum-Based Chemotherapy and Bevacizumab as First Line Treatment in Patients With Recurrent, Persistent or Metastatic Cervical Cancer
Brief Title: Efficacy and Safety of BCD-100 (Anti-PD-1) in Combination With Platinum-Based Chemotherapy and Bevacizumab in Patients With Recurrent, Persistent or Metastatic Cervical Cancer (CAESURA)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCD-100-4/CAESURA
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Cervical Cancer; Cervical Cancer Metastatic; Cervical Cancer Recurrent
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Bevacizumab; Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCD-100 (Experimental): BCD-100 mg/kg Q3W
  Interventions: Biological: BCD-100; Biological: Bevacizumab; Drug: Paclitaxel; Drug: Cisplatin (or carboplatin)

INTERVENTIONS:
Biological: BCD-100 — Anti-PD-1 monoclonal antibody, IV infusion
Biological: Bevacizumab — IV infusion
Drug: Paclitaxel — IV infusion
Drug: Cisplatin (or carboplatin) — IV infusion

SUMMARY:
This is a multicenter, open-label, single-arm study of efficacy, safety and pharmacokinetics of BCD-100 (JSC BIOCAD, Russia) in combination with platinum-based chemotherapy and bevacizumab as first-line treatment in patients with recurrent/persistent or metastatic cervical cancer.

DETAILED DESCRIPTION:
The study will be conducted in two stages. At the first stage patients will receive up to 6 cycles of BCD-100 in combination with platinum-based chemotherapy and bevacizumab or until unacceptable toxicity or disease progression. Patients who have demonstrated a positive antitumor effect (stabilization of the disease, partial or complete response) and who have no signs of unacceptable toxicity could continue to receive up to 12 cycles of maintenance therapy of BCD-100 in combination with bevacizumab or until unacceptable toxicity or disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form and the subject's ability to follow the Protocol requirements;
2. Age: 18 years and older at the signing of the informed consent;
3. Histologically verified (documented) adenomatous, adenosquamous, or squamous cervical cancer;
4. Newly diagnosed metastatic cervical cancer or recurrent/persistent cervical cancer;
5. Availability of archival histological tumor material (paraffin blocks) or consent to biopsy;
6. ECOG performance status of 0 or 1;
7. At least one RESICT 1.1-defined measurable target lesion confirmed by an independent review;
8. Patients with reproductive potential must agree to practice acceptable methods of birth control throughout the entire trial period, starting from signing the informed consent and up to 24 weeks after the last dose of investigational product.

Exclusion Criteria:

1. Indications for radical therapy (surgical or radiotherapy);
2. Prior systemic treatment for recurrent, secondarily progressive or initially metastatic disease;
3. Chemotherapy, and / or radiation therapy, and / or chemo-radiation therapy for early stages of cervical cancer with disease progression / recurrence earlier than 6 months after the end of therapy;
4. Patients with severe concomitant factors or the effects of their treatment (hemorrhage, perforation, fistula);
5. Central nervous system (CNS) metastases;
6. Concomitant diseases or conditions which pose a risk of AE development during study treatment:

   1. uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg;
   2. stable angina functional class III-IV;
   3. unstable angina or myocardial infarction less than 6 months prior to randomization;
   4. NYHA Grade III-IV congestive heart failure;
   5. atopic asthma, Stage III-IV COPD, angioedema;
   6. severe respiratory failure;
   7. any other diseases which pose unacceptable risk of AE development during study treatment in Investigator's opinion;
7. Active or known or suspected autoimmune disease (subjects with Type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, or skin disorders (vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll);
8. Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days prior to randomization;
9. Established diagnosis of coagulopathy and / or clinically significant bleeding, including nasal bleeding;
10. The need for regular intake of anticoagulants, antiplatelet agents, platelet function inhibitors, or their course application less than 1 month before being included in the study;
11. Hematologic disorders: neutrophils <1500/mcl or platelets <100 000/mcl or hemoglobin <90 g/l;
12. Renal disorders: creatinine ≥ 1.5 x UNL;
13. Hepatic disorders: bilirubin ≥ 1.5 x UNL (excluding Gilbert's syndrome if bilirubin < 50 µmol/l) or AST/ALT ≥ 3 x UNL (excluding subjects with liver metastases if AST/ALT < 5 x UNL) or alkaline phosphatase ≥ 5 x UNL;
14. Any anti-cancer therapy less than 28 days prior to randomization;
15. Previous use of PD-1/PD-L1/PD-L2/CTLA-4 agent;
16. Previous use of VEGF/VEGFR inhibitors, including bevacizumab, ramucirumab, aflibercept and tyrosine kinase inhibitors;
17. Concomitant cancer (except for cervical carcinoma in situ after radical surgery or basal cell/ squamous cell carcinoma after radical surgery);
18. Clinically significant (≥2 degree) peripheral neuropathy or hearing impairment;
19. Any condition that prevents a patient from following the Protocol procedures (dementia, neurological or mental disorders, drug/alcohol abuse, etc.);
20. Simultaneous participation in other clinical trials , participation in other clinical trials within 30 days prior to the first dose of the investigational product;
21. Acute infection or the acute phase of chronic infection within 28 days prior the first dose of the investigational product;
22. Active HBV/HCV/HIV infection, active syphilis;
23. Patients unable to receive an IV infusions;
24. Patients unable to receive an IV contrast agent;
25. Hypersensitivity to any of the components of BCD-100, bevacizumab, paclitaxel, cisplatin (or carboplatin);
26. Life expectancy less than 6 months;
27. Significant adverse events (AE) of previous therapy excluding chronic and/or irreversible events which cannot affect study drug safety evaluation (e.g. alopecia);
28. Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2018-12-25 (Actual); Primary Completion 2020-07-07 (Estimated); Study Completion 2020-07-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  ORR is defined as the percentage of the participants in the mITT population who have a Complete Response or a Partial Response. The ORR will be assessed by a blind independent central reviewer per RECIST 1.1 and iRECIST.

SECONDARY OUTCOMES:
Median Progression-free Survival (PFS) | 1 year
1-year Progression-free Survival (PFS) | 1 year
1-year Overall Survival (OS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roman A Ivanov, PhD, Study Director — Vice President R&D, JSC BIOCAD
Locations (24):
- Russia (24):
  - City Hospital No. 5, Barnaul, Altayskiy Kray
  - Arkhangelsk Clinical Oncology Dispensary, Arkhangelsk, Arkhangelskaya oblast
  - Chelyabinsk Regional Clinical Center for Oncology and Nuclear Medicine, Chelyabinsk, Chelyabinsk Oblast
  - National Medical Radiology Research Center, Obninsk, Kaluga Oblast
  - Clinical Oncologic Dispensary No. 1, Krasnodar, Krasnodar Kari
  - Krasnoyarsk Regional Clinical Oncological Dispensary named after A.I. Kryzhanovsky, Krasnoyarsk, Krasnoyarsk Krai
  - Murmansk Regional Clinical Hospital named after P.A. Bayandina, Murmansk, Murmansk Oblast
  - Clinical Oncology Dispensary, Omsk, Omsk Oblast
  - Republican Oncology Center, Saransk, Respublika Mordoviya
  - N.N. Petrov National Medical Research Center of Oncology (2), Saint Petersburg, Sankt-Peterburg
  - LLC "New Clinic", Pyatigorsk, Stavropol Kray
  - Stavropol Regional Clinical Oncology Center, Stavropol, Stavropol Kray
  - Sverdlovsk Regional Oncology Center, Yekaterinburg, Sverdlovsk Oblast
  - Republican Clinical Oncology Cente, Kazan', Tatarstan Republic
  - Regional Clinical Oncology Hospital, Yaroslavl, Yaroslavl Oblast
  - Moscow Clinical Scientific and Practical Center named A.S. Loginova, Moscow
  - N.N. Blokhin National Medical Research Center of Oncology (2), Moscow
  - N.N. Blokhin National Medical Research Center of Oncology, Moscow
  - JSC "Medsi Group of Companies", Moscow
  - Moscow City Oncology Hospital No. 62, Moscow
  - JSC "Modern Medical Technologies", Saint Petersburg
  - LLC "AB Medical Group", Saint Petersburg
  - N.N. Petrov National Medical Research Center of Oncology, Saint Petersburg
  - Saint-Petersburg Petersburg Clinical Scientific and Practical Center for Specialized Types of Medical Care (Oncological), Saint Petersburg

IPD SHARING:
Plan to Share IPD: No